CLINICAL TRIAL: NCT04868929
Title: The Brain Activation During Motor Execution, Motor Imagery, Action Observation, and Mirror Visual Feedback in Healthy Adults
Brief Title: The Brain Activation During Different Motor Patterns in Healthy Adults
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202102037RINA
Record Dates: First submitted 2021-04-25; First posted 2021-05-03 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-06

CONDITIONS: Neurosciences
Keywords: brain activation; near infrared spectroscopy; motor imagery; action observation; mirror visual feedback

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to investigate the brain activation during different motor patterns, including motor execution (ME), motor imagery (MI), action observation (AO) and mirror visual feedback (MVF). In addition, the relations between brain activation and motor performance will also be explored. This study includes two parts, which are upper limb and lower limb part. While executing all the tasks, brain activation in primary motor cortex(M1), premotor cortex(PMC), and supplementary motor cortex(SMA) will be monitored by functional near-infrared spectroscopy. One-way ANOVA with repeated measure will be used to detect the differences of brain activation level between each mode. Pearson correlation coefficient will be used to determine the relations of brain activation and motor performance.

DETAILED DESCRIPTION:
In upper limb part, subjects will be instructed to execute functional reaching task in ME, MI, AO, and MVF mode. During ME mode, motor performance including maximum speed, maximum acceleration, and jerk will be collected simultaneously. In the lower limb part, subjects will be instructed to walking over ground in ME, MI, and AO mode. During ME mode, the temporal and spatial gait parameters, including speed, stride time, cadence, and stride length will be collected.

ELIGIBILITY:
* Inclusion Criteria

  1. Age between 20 to 30 years.
  2. Right-handed.
  3. Ability to walk 30 meters independently without an assistive device.
  4. No neurogical, cardiopulmonary, or muscle diseases that might interfere with the experiment.
  5. Mini-Mental State Examination (MMSE) score greater than 24.
* Exclusion Criteria 1. Physiological condition is unstable.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population in this study are heathly adults.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-08-07 (Actual); Study Completion 2022-08-07 (Actual)

PRIMARY OUTCOMES:
Brain activities over primary motor cortex | Day 1
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over premotor cortex | Day 1
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over supplementary motor area | Day 1
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.

SECONDARY OUTCOMES:
Motor performance of upper limb -maximum speed | Day 1
  cm/s
Motor performance of upper limb -maximum acceleration | Day 1
  cm/s^2
Motor performance of upper limb - jerk | Day 1
  cm/s^3
Motor performance of lower limb - gait speed | Day 1
  cm/s
Motor performance of lower limb - cadence | Day 1
  steps
Motor performance of lower limb - stride time | Day 1
  second
Motor performance of lower limb - stride length | Day 1
  cm

CONTACTS AND LOCATIONS:
Overall Officials: Yanci Liu, PHD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan